CLINICAL TRIAL: NCT00505778
Title: A Multi-center, Investigator-blinded, Randomized, 12-month, Parallel-group, Non-inferiority Study to Compare the Efficacy of 1.6 to 2.4 g Asacol® Therapy QD Versus Divided Dose (BID) in the Maintenance of Remission of Ulcerative Colitis
Brief Title: A Comparison of Once a Day Dose Compared to 2 Doses/Day
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Warner Chilcott (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2007021
Record Dates: First submitted 2007-07-20; First posted 2007-07-23 (Estimated); Results first posted 2011-05-12 (Estimated); Last update posted 2013-04-22 (Estimated); Status verified 2013-04

CONDITIONS: Ulcerative Colitis
MeSH Terms: conditions — Colitis, Ulcerative

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Mesalamine (Asacol) Once-Daily (Active Comparator): an oral, once daily (QD) mesalamine regimen (1.6 - 2.4 g/day)
  Interventions: Drug: Mesalamine Once-Daily
- Mesalamine (Asacol) Twice-Daily (Active Comparator): an oral, twice daily (BID) mesalamine regimen (1.6 - 2.4 g/day)
  Interventions: Drug: Mesalamine Twice-Daily

INTERVENTIONS:
Drug: Mesalamine Once-Daily — Mesalamine tablets, 1.6-2.4 g/day taken orally once a day for 52 weeks
  Other Names: Asacol QD
  Arms: Mesalamine (Asacol) Once-Daily
Drug: Mesalamine Twice-Daily — Mesalamine tablets, 1.6-2.4 g/day, taken twice daily for 52 weeks
  Other Names: Asacol BID
  Arms: Mesalamine (Asacol) Twice-Daily

SUMMARY:
The purpose of this study is to compare the efficacy in maintaining remission of ulcerative colitis between a once daily (QD) Asacol regimen and a divided, twice daily (BID) Asacol dosing regimen.

DETAILED DESCRIPTION:
Currently, in the US, Asacol therapy is indicated in divided doses for the maintenance of remission of ulcerative colitis at 1.6 g/day. A once daily dose is potentially beneficial to patients and physicians alike. This study will answer the following questions about once daily dosing: (1) does efficacy differ between once daily and twice daily dosing, (2) do patients prefer a once daily dosing regimen, and (3) is compliance better? This study will confirm whether there are benefits to once daily dosing beyond increased convenience. In order to understand how the QD regimen compares to BID in a "real life" practice setting, the patient will remain on the total daily dose of Asacol (1.6 g/day to 2.4 g/day) on which they were maintained in remission, but will be assigned to either a QD or BID regimen. This is an investigator-blinded study.

ELIGIBILITY:
Inclusion Criteria:

* Documented history of ulcerative colitis that has been successfully maintained in remission for at least 3 months prior to study entry
* At least one flare in the past 18 months
* Utilizing a stable maintenance dose of oral Asacol of 1.6 g/day up to 2.4 g/day (stable dose is defined as the same dose for the past 3 months)
* Females must be postmenopausal or surgically sterile or have a negative urine pregnancy test and practice acceptable contraception

Exclusion Criteria:

* History of or current renal disease
* History of hepatic disease
* History of allergy or hypersensitivity to salicylates, aminosalicylates
* Treatment with immunomodulatory therapy, biologic therapy or corticosteroids within 90 days of screening
* Received any antidiarrheals, antispasmodics, or antibiotic within 1 month of screening

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1027 (Actual)
Dates: Start 2007-07; Primary Completion 2009-07 (Actual); Study Completion 2009-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tom G Todaro, MD, Study Director — Procter and Gamble
Locations (217):
- United States (208):
  - Research Facility, Athens, Alabama
  - Research Facility, Birmingham, Alabama
  - Research Facility, Dothan, Alabama
  - Research Facility, Phoenix, Arizona
  - Research Facility, Scottsdale, Arizona
  - Research Facility, Tucson, Arizona
  - Research Facility, Tuscon, Arizona
  - Research Facility, Little Rock, Arkansas
  - Research Facility, Lowell, Arkansas
  - Research Facility, Anaheim, California
  - Research Facility, Beverly Hills, California
  - Research Facility, Chico, California
  - Research Facility, Encinitas, California
  - Research Facility, Folsom, California
  - Research Facility, La Mesa, California
  - Research Facility, Lancaster, California
  - Research Facility, Long Beach, California
  - Research Facility, Los Angeles, California
  - Research Facility, Madera, California
  - Research Facility, Merced, California
  - Research Facility, Mission Hills, California
  - Research Facility, Monterey, California
  - Research Facility, Murrieta, California
  - Research Facility, Oakland, California
  - Research Facility, Orange, California
  - Research Facility, Palm Springs, California
  - Research Facility, San Carlos, California
  - Research Facility, San Diego, California
  - Research Facility, San Francisco, California
  - Research Facility, Torrance, California
  - Research Facility, Upland, California
  - Research Facility, Englewood, Colorado
  - Research Facility, Golden, Colorado
  - Research Facility, Lafayette, Colorado
  - Research Facility, Pueblo, Colorado
  - Research Facility, Hartford, Connecticut
  - Research Facility, Meriden, Connecticut
  - Research Facility, New Haven, Connecticut
  - Research Facility, Norwalk, Connecticut
  - Research Facility, Torrington, Connecticut
  - Research Facility, Washington D.C., District of Columbia
  - Research Facility, Aventura, Florida
  - Research Facility, Fort Lauderdale, Florida
  - Research Facility, Gainesville, Florida
  - Research Facility, Hollywood, Florida
  - Research Facility, Jacksonville, Florida
  - Research Facility, Largo, Florida
  - Research Facility, Maitland, Florida
  - Research Facility, Naples, Florida
  - Research Facility, New Port Richey, Florida
  - Research Facility, North Miami Beach, Florida
  - Research Facility, Orlando, Florida
  - Research Facility, Palm Harbor, Florida
  - Research Facility, Port Orange, Florida
  - Research Facility, St. Petersburg, Florida
  - Research Facility, Tallahassee, Florida
  - Research Facility, Tampa, Florida
  - Research Facility, Trinity, Florida
  - Research Facility, Winter Park, Florida
  - Research Facility, Zephyrhills, Florida
  - Research Facility, Atlanta, Georgia
  - Research Facility, Columbus, Georgia
  - Research Facility, Decatur, Georgia
  - Research Facility, Marietta, Georgia
  - Research Facility, Newnan, Georgia
  - Research Facility, Savannah, Georgia
  - Research Facility, Boise, Idaho
  - Research Facility, Idaho Falls, Idaho
  - Research Facility, Arlington Heights, Illinois
  - Research Facility, Berwyn, Illinois
  - Research Facility, Chicago, Illinois
  - Research Facility, Elgin, Illinois
  - Research Facility, Highland Park, Illinois
  - Research Facility, Hoffman Estates, Illinois
  - Research Facility, Homewood, Illinois
  - Research Facility, Lake Barrington, Illinois
  - Research Facility, Oak Lawn, Illinois
  - Research Facility, Peoria, Illinois
  - Research Facility, Urbana, Illinois
  - Research Facility, Anderson, Indiana
  - Research Facility, Bloomington, Indiana
  - Research Facility, Indianapolis, Indiana
  - Research Facility, South Bend, Indiana
  - Research Facility, Clive, Iowa
  - Research Facility, Davenport, Iowa
  - Research Facility, Waterloo, Iowa
  - Research Facility, Pratt, Kansas
  - Research Facility, Topeka, Kansas
  - Research Site, Whichita, Kansas
  - Research Facility, Bowling Green, Kentucky
  - Research Facility, Louisville, Kentucky
  - Research Facility, Alexandria, Louisiana
  - Research Facility, Lafayette, Louisiana
  - Research Facility, Metairie, Louisiana
  - Research Facility, Monroe, Louisiana
  - Research Facility, Shreveport, Louisiana
  - Research Facility, Bangor, Maine
  - Research Facility, Chevy Chase, Maryland
  - Research Facility, College Park, Maryland
  - Research Facility, Greenbelt, Maryland
  - Research Facility, Hagerstown, Maryland
  - Research Facility, Hollywood, Maryland
  - Research Facility, Lutherville, Maryland
  - Research Facility, Reisterstown, Maryland
  - Research Facility, Rockville, Maryland
  - Research Facility, Boston, Massachusetts
  - Research Facility, Braintree, Massachusetts
  - Research Facility, Southbridge, Massachusetts
  - Research Facility, Chesterfield, Michigan
  - Research Facility, Detroit, Michigan
  - Research Facility, Kalamazoo, Michigan
  - Research Facility, Troy, Michigan
  - Research Facility, West Bloomfied, Michigan
  - Research Facility, Wyoming, Michigan
  - Research Facility, Rochester, Minnesota
  - Research Facility, Tupelo, Mississippi
  - Research Facility, Cape Girardeau, Missouri
  - Research Facility, Columbia, Missouri
  - Research Facility, Jefferson City, Missouri
  - Research Facility, Mexico, Missouri
  - Research Facility, St Louis, Missouri
  - Research Facility, Las Vegas, Nevada
  - Research Facility, Somersworth, New Hampshire
  - Research Facility, Camden, New Jersey
  - Research Facility, Cedar Knolls, New Jersey
  - Research Facility, Egg Harbor, New Jersey
  - Research Site, Hackensack, New Jersey
  - Research Facility, Ocean City, New Jersey
  - Research Facility, South Plainfield, New Jersey
  - Research Facility, Albuquerque, New Mexico
  - Research Facility, Babylon, New York
  - Research Facility, Binghamton, New York
  - Research Facility, Brooklyn, New York
  - Research Facility, Cheektowaga, New York
  - Research Facility, Cortland, New York
  - Research Facility, Forest Hills, New York
  - Research Facility, Garden City, New York
  - Research Facility, Great Neck, New York
  - Research Facility, Lake Success, New York
  - Research Facility, New York, New York
  - Research Facility, Pittsford, New York
  - Research Facility, Port Jefferson Station, New York
  - Research Facility, Rochester, New York
  - Research Facility, Boone, North Carolina
  - Research Facility, Charlotte, North Carolina
  - Research Facility, Greensboro, North Carolina
  - Research Facility, Greenville, North Carolina
  - Research Facility, Jacksonville, North Carolina
  - Research Facility, Kinston, North Carolina
  - Research Facility, Morganton, North Carolina
  - Research Facility, Mount Airy, North Carolina
  - Research Facility, New Bern, North Carolina
  - Research Facility, Pinehurst, North Carolina
  - Research Facility, Raleigh, North Carolina
  - Research Facility, Wilmington, North Carolina
  - Research Facility, Bismarck, North Dakota
  - Research Facility, Akron, Ohio
  - Research Facility, Canton, Ohio
  - Research Facility, Cincinnati, Ohio
  - Research Facility, Cleveland, Ohio
  - Research Facility, Dayton, Ohio
  - Research Facility, Mentor, Ohio
  - Research Facility, Toledo, Ohio
  - Research Facility, Westlake, Ohio
  - Research Facility, Tulsa, Oklahoma
  - Research Facility, Portland, Oregon
  - Research Facility, Allentown, Pennsylvania
  - Research Facility, Beaver Falls, Pennsylvania
  - Research Facility, Clairton, Pennsylvania
  - Research Facility, Indiana, Pennsylvania
  - Research Facility, Lancaster, Pennsylvania
  - Research Facility, Philadelphia, Pennsylvania
  - Research Facility, Phoenixville, Pennsylvania
  - Research Facility, Pittsburgh, Pennsylvania
  - Research Facility, Sewickley, Pennsylvania
  - Research Facility, Souderton, Pennsylvania
  - Research Facility, Uniontown, Pennsylvania
  - Research Facility, Warwick, Rhode Island
  - Research Facility, Columbia, South Carolina
  - Research Facility, Greer, South Carolina
  - Research Facility, Jackson, Tennessee
  - Research Facility, Memphis, Tennessee
  - Research Facility, Morristown, Tennessee
  - Research Facility, Amarillo, Texas
  - Research Facility, Fort Worth, Texas
  - Research Facility, Greenville, Texas
  - Research Facility, Houston, Texas
  - Research Facility, Lewisville, Texas
  - Research Facility, Longview, Texas
  - Research Facility, Odessa, Texas
  - Research Facility, Pasadena, Texas
  - Research Facility, Plano, Texas
  - Research Facility, San Antonio, Texas
  - Research Facility, Ogden, Utah
  - Research Facility, Salt Lake City, Utah
  - Research Facility, West Valley City, Utah
  - Research Facility, Alexandria, Virginia
  - Research Facility, Chesapeake, Virginia
  - Research Facility, Fairfax, Virginia
  - Research Facility, Norfolk, Virginia
  - Research Facility, Virginia Beach, Virginia
  - Research Facility, Winchester, Virginia
  - Research Facility, Seattle, Washington
  - Research Facility, Spokane, Washington
  - Research Facility, Tacoma, Washington
  - Research Facility, Wenatchee, Washington
  - Research Facility, Milwaukee, Wisconsin
  - Research Facility, Monroe, Wisconsin
- Canada (7):
  - Research Facility, Abbotsford, British Columbia
  - Research Facility, Guelph, Ontario
  - Research Facility, Hamilton, Ontario
  - Research Facility, Ottawa, Ontario
  - Research Facility, Toronto, Ontario
  - Research Facility, Montreal, Quebec
  - Research Facility, Québec, Quebec
- Puerto Rico (2):
  - Research Facility, Ponce
  - Research Facility, San Juan

REFERENCES:
- [Derived] Sandborn WJ, Korzenik J, Lashner B, Leighton JA, Mahadevan U, Marion JF, Safdi M, Sninsky CA, Patel RM, Friedenberg KA, Dunnmon P, Ramsey D, Kane S. Once-daily dosing of delayed-release oral mesalamine (400-mg tablet) is as effective as twice-daily dosing for maintenance of remission of ulcerative colitis. Gastroenterology. 2010 Apr;138(4):1286-96, 1296.e1-3. doi: 10.1053/j.gastro.2009.12.054. Epub 2010 Jan 11. PMID 20064514

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Enrollment began 9 Aug 2007
Groups:
- Mesalamine Once-Daily: an oral, once daily (QD) mesalamine regimen (1.6 - 2.4 g/day)
- Mesalamine Twice-Daily: an oral, twice daily (BID) mesalamine regimen (1.6 - 2.4 g/day)
Period: Overall Study
Arm/Group | Mesalamine Once-Daily | Mesalamine Twice-Daily
Started | 514 | 513
Intent to Treat (ITT) Population | 512 | 511
Completed | 380 | 378
Not Completed | 134 | 135
Not completed — Adverse Event | 2 | 7
Not completed — Physician Decision | 8 | 14
Not completed — Lost to Follow-up | 17 | 23
Not completed — Unable to Meet Protocol Criteria | 4 | 1
Not completed — Protocol Violation | 7 | 9
Not completed — Withdrawal by Subject | 29 | 14
Not completed — Relapse | 65 | 65
Not completed — Took No Study Drug | 2 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Mesalamine Once-Daily | Mesalamine Twice-Daily | Total
Number analyzed (Participants) | 514 | 513 | 1027
Age, Customized [Number; unit: Participants] — ITT Population
  Participants
    < 65 years old | 409 | 414 | 823
    > = 65 years old | 103 | 97 | 200
Gender [Number; unit: participants] — ITT Population
  participants
    Female | 261 | 268 | 529
    Male | 251 | 243 | 494
Region of Enrollment [Number; unit: participants] — ITT Population
  participants
    Canada | 6 | 8 | 14
    United States | 506 | 503 | 1009

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Patients Remaining in Remission at Month 6, ITT Population, Determined by the Simple Clinical Colitis Activity Index (SCCAI)
Description: Remission defined as SCCAI <5. Simple Clinical Colitis Activity Index: minimum score 0, maximum score 19, reflects disease activity over the 24 hours prior to completion. Composite Score: bowel frequency (day, 0-3) (night, 0-2), defecation urgency (0-3), blood in stool (0-3), general well being (0-4), extracolonic features (arthritis, pyoderma gangrenosum, erythema nodosum, uveitis - 1 per manifestation).
Time Frame: 6 months
Population: ITT Population
Measure: Number; unit: Percentage of Participants
Arm/Group | Mesalamine Once-Daily | Mesalamine Twice-Daily
Number analyzed (Participants) | 512 | 511
Percentage of Participants | 90.5 | 91.8
Statistical Analysis 1: Comparison: Mesalamine Once-Daily vs Mesalamine Twice-Daily; Assumed true remission rate is 70% with no difference in remission rates between QD and BID dosing.The non-inferiority margin used in hypothesis testing was set to 10%; Test type: Non-Inferiority or Equivalence — To establish non-inferiority for primary efficacy variable at 2-sided upper confidence bound of 95% with 90% power, 442 patients per treatment group were required to be analyzable for primary efficacy analysis. Assuming 10% enrolled would not be analyzable, 1000 patients would be enrolled. If the 95% confidence interval's upper bound interval for the difference between the Asacol BID and Asacol QD group is <10%, then non-inferiority of Asacol QD is claimed; p = 0.5016, Cochran-Mantel-Haenszel; Stratified by prior Asacol dose Category; BID-QD Difference in Remission Rates = 1.3, 95% CI 2-sided [-2.3 to 4.9]

2. Secondary Outcome: Percentage of Patients Remaining in Remission at Month 3, ITT Population
Description: Remission defined as SCCAI < 5. Simple Clinical Colitis Activity Index: minimum score 0, maximum score 19, reflects disease activity over the 24 hours prior to completion. Composite Score: bowel frequency (day, 0-3) (night, 0-2), defecation urgency (0-3), blood in stool (0-3), general well being (0-4), extracolonic features (arthritis, pyoderma gangrenosum, erythema nodosum, uveitis - 1 per manifestation).
Time Frame: 3 months
Population: ITT Population
Measure: Number; unit: Percentage of Participants
Arm/Group | Mesalamine Once-Daily | Mesalamine Twice-Daily
Number analyzed (Participants) | 512 | 511
Percentage of Participants | 94.8 | 95.6
Statistical Analysis 1: Comparison: Mesalamine Once-Daily vs Mesalamine Twice-Daily; [analysis description as in outcome 1, analysis 1]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.5426, Cochran-Mantel-Haenszel; Stratified by prior Asacol dose Category; BID-QD Difference in Remission Rates = 0.8, 95% CI 2-sided [-1.8 to 3.5]

3. Secondary Outcome: Percentage of Patients Remaining in Remission at Month 12, ITT Population
Description: Remission defined as SCCAI score < 5. Simple Clinical Colitis Activity Index: minimum score 0, maximum score 19, reflects disease activity over the 24 hours prior to completion. Composite Score: bowel frequency (day, 0-3) (night, 0-2), defecation urgency (0-3), blood in stool (0-3), general well being (0-4), extracolonic features (arthritis, pyoderma gangrenosum, erythema nodosum, uveitis - 1 per manifestation).
Time Frame: 12 months
Population: ITT Population
Measure: Number; unit: Percentage of Participants
Arm/Group | Mesalamine Once-Daily | Mesalamine Twice-Daily
Number analyzed (Participants) | 512 | 511
Percentage of Participants | 85.4 | 85.4
Statistical Analysis 1: Comparison: Mesalamine Once-Daily vs Mesalamine Twice-Daily; [analysis description as in outcome 1, analysis 1]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.9770, Cochran-Mantel-Haenszel; Stratified by prior Asacol dose Category; BID-QD Difference in Remission Rates = 0.0, 95% CI 2-sided [-4.6 to 4.7]

4. Secondary Outcome: Number of Subjects Who Relapse/Flare Within 6 Months, ITT Population
Description: Relapse/flare is defined as SCCAI >= 5. Simple Clinical Colitis Activity Index: minimum score 0, maximum score 19, reflects disease activity over the 24 hours prior to completion. Composite Score: bowel frequency (day, 0-3) (night, 0-2), defecation urgency (0-3), blood in stool (0-3), general well being (0-4), extracolonic features (arthritis, pyoderma gangrenosum, erythema nodosum, uveitis - 1 per manifestation).
Time Frame: 6 months
Population: ITT Population
Measure: Number; unit: Participants
Arm/Group | Mesalamine Once-Daily | Mesalamine Twice-Daily
Number analyzed (Participants) | 512 | 511
Participants | 45 | 39
Statistical Analysis 1: Comparison: Mesalamine Once-Daily vs Mesalamine Twice-Daily; Test type: Superiority or Other; p = 0.4726, Log Rank; Stratified by prior Asacol dose Category; Hazard Ratio (HR) = 1.170, 95% CI 2-sided [0.762 to 1.796]

5. Secondary Outcome: Total MARS (Medication Adherence Report Scale) Questionnaire Scores, ITT Population, Month 6
Description: MARS: Composite score for the following statements: I change how many times per day I take my medicine, I forget to use it, I stop taking it for a while, I only use it when I am having active symptoms, I decide to miss out on a dose, I take less than instructed, I take more than instructed, I avoid using it if I can, I use it regularly every day (reverse scored): 5-never, 4-rarely, 3-sometimes, 2-often, 1-very often. Minimum score 9, maximum score 45.
Time Frame: 6 months
Population: ITT Population
Measure: Mean (Standard Error); unit: MARS Score
Arm/Group | Mesalamine Once-Daily | Mesalamine Twice-Daily
Number analyzed (Participants) | 512 | 511
MARS Score | 42.3 (0.23) | 41.8 (0.24)
Statistical Analysis 1: Comparison: Mesalamine Once-Daily vs Mesalamine Twice-Daily; Test type: Superiority or Other; p = 0.1753, ANOVA; ANOVA with prior Asacol dose category as factor; Difference BID-QD in Least Square Mean = -0.45, 95% CI 2-sided [-1.09 to 0.20]

6. Secondary Outcome: Percentage of Participants Indicating Ulcerative Colitis in Remission (Patient Defined Remission Index), ITT Population, Month 6
Description: Is your ulcerative colitis in remission (not active)? Y/N
Time Frame: 6 months
Population: ITT Population
Measure: Number; unit: Percentage of Participants
Arm/Group | Mesalamine Once-Daily | Mesalamine Twice-Daily
Number analyzed (Participants) | 512 | 511
Percentage of Participants | 83.1 | 86.6
Statistical Analysis 1: Comparison: Mesalamine Once-Daily vs Mesalamine Twice-Daily; [analysis description as in outcome 1, analysis 1]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.1557, Cochran-Mantel-Haenszel; Stratified by prior Asacol dose Category; Difference BID-QD Remission Rates = 3.6, 95% CI 2-sided [-1.3 to 8.5]

ADVERSE EVENTS:
Time Frame: 12 months
Description: ITT Population, Only Immediately Reportable Events (SAEs or withdrawal due to AEs) collected for this study. Data collected between 9 Aug 2007 and 29 Jul 2009.
Arm/Group | Mesalamine Once-Daily | Mesalamine Twice-Daily
Serious Adverse Events (participants affected / at risk) | 18/512 | 9/511
Other Adverse Events (participants affected / at risk) | 0/512 | 0/511
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Mesalamine Once-Daily (N=512) | Mesalamine Twice-Daily (N=511)
Abdominal Pain (Gastrointestinal disorders) | 0 | 1
Ascites (Gastrointestinal disorders) | 0 | 1
Constipation (Gastrointestinal disorders) | 0 | 1
Rectal Haemorrhage (Gastrointestinal disorders) | 0 | 1
Anal fistula (Gastrointestinal disorders) | 1 | 0
Breast Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Oesophageal Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Small Cell Lung Cancer Metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Renal Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Thyroid Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Uterine Leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Cardiomyopathy (Cardiac disorders) | 0 | 1
Coronary Artery Disease (Cardiac disorders) | 0 | 1
Atrial Fibrillation (Cardiac disorders) | 1 | 0
Cardiac Failure Congestive (Cardiac disorders) | 1 | 0
Myocardial Infarcation (Cardiac disorders) | 1 | 0
Renal Failure Acute (Renal and urinary disorders) | 0 | 2
Dehydration (Metabolism and nutrition disorders) | 0 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 0
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Haemothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Deep Vein Thrombosis (Vascular disorders) | 0 | 1
Hypertension (Vascular disorders) | 1 | 0
Thrombophlebitis (Vascular disorders) | 1 | 0
Cholangitis (Hepatobiliary disorders) | 1 | 0
Cholelithiasis (Hepatobiliary disorders) | 2 | 0
Jaundice Cholestatic (Hepatobiliary disorders) | 1 | 0
Appendicitis (Infections and infestations) | 2 | 0
Diverticulitis (Infections and infestations) | 1 | 0
Clavicle Fracture (Injury, poisoning and procedural complications) | 1 | 0
Rib Fracture (Injury, poisoning and procedural complications) | 1 | 0
Spinal Compression Fracture (Injury, poisoning and procedural complications) | 1 | 0
Altered State of Consciousness (Nervous system disorders) | 1 | 0
Convulsion (Nervous system disorders) | 1 | 0
Transient Ischaemic Attack (Nervous system disorders) | 1 | 0
Chest Pain (General disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less